CLINICAL TRIAL: NCT03801018
Title: Gamete Donation Conception and Disclosure to Children : Towards an Evaluation of the Practices
Brief Title: Gamete Donation Conception and Disclosure to Children : Towards an Evaluation of the Practices (AMP)
Acronym: AMP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-53
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-12

CONDITIONS: Assisted Reproductive Techniques
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents who have used the donation of gametes
  Interventions: Other: Questionnary and Interviews
- Children born of gametes donation
  Interventions: Other: Questionnary and Interviews

INTERVENTIONS:
Other: Questionnary and Interviews — An internet platform dedicated to the anonymous survey will be set up by the communication department and the digital System Department of the promoter Public assistance hospitals in Marseille, the data Processing manager. It would deplore anonymous questionnaires accessible from a dedicated web page. People will therefore respond to a national survey on the basis of volunteering and anonymity.
  Interviews, lasting one to two hours, will be fully transcribed and processed anonymously.
  The interviews will seek to collect data on the modalities, conditions and effects of the circulation (or retention) of information on the use of donation, throughout the lives of individuals and families, in a cross-analysis of Viewpoints of parents and people born of donation.

SUMMARY:
Assisted reproductive techniques (ART) is very framed in France by principles initially stated by the french CECOS Federation of (Centre d'Etude et de Conservation des Oeufs et du Sperme) and then included in the bioethic law. Since 1973, more than 50 000 births have been achieved through sperm donation, and the investigators have little knowledge of what information parents pass on to their children about how they have conceived. However, it is accepted that the secrecy about the use of donated gametes has negative consequences.

The investigators propose an original project never initiated in France, to evaluate at the national level the disclosure to the people conceived using donated gametes, thanks to an interdisciplinary research crossing medical approach (biology, psychology) and social sciences (anthropology, sociology). It uses a quantitave and qualitative approach relying on one hand on online questionnaires and on the other hand on semi-structured interviews, aimed at parent who have used ART with donated gametes and people conceived using donated gametes. This dual approach will outline broad trends in sharing information about the use of donated gametes, explore in depth the motivation of parental choices for information, and better understand the family and biographical dynamics associated with information sharing or its absence. Moreover, this project will lead to evaluate the way in which the parents received the messages of the professionnals involved in ART with donation gametes, in terms of disclosure to offspring.

The conclusions will highlight the most important elements that will be useful to the professionnals involved in gamete donation to help them improve their practices upstream, during, and after the completion of the ART with gamete donation.

ELIGIBILITY:
Inclusion Criteria:

For the parents :

* Parents of children from sperm donation
* Parents of children from oocyte donation
* Major people
* Parents who have benefited from taking over in France or taking charge in a foreign country, in a legal framework different from ours
* People who gave their non-opposition

For the childs :

* Person born by sperm donation
* Person born by Egg donation
* Major person
* Person who gave their non-opposition

Exclusion Criteria:

* Minor person
* No one who has used the amp or anyone who is not from an amp with gamete donation.
* People who have not expressed their non-opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents of children from gametes donation Person born by gametes donation
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-01-06 (Estimated); Study Completion 2021-01-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate, for parents who have informed their child, how and when the information was circulated. | 2 Years
  An internet platform dedicated to the anonymous survey will be set up by the communication department and the digital System Department of the promoter Public assistance hospitals in Marseille.
  A first questionnaire will be for the parents, the second questionnaire will be for people born through a donation. They will include closed questions, drop-down menus and rare open questions. The succession of questions will be studied in order to check the consistency of the answers. Replies to the questionnaires can be extracted anonymously.
  The interviews will seek to collect data on the modalities, conditions and effects of the circulation (or retention) of information on the use of donation, throughout the lives of individuals and families, in a cross-analysis of Viewpoints of parents and people born of Don.
  A cross-analysis of quantitative and qualitative data will be carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Olivier Arnaud, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- service de Biologie de la Reproduction-CECOS, Marseille, Marseille Cedex 5, France